CLINICAL TRIAL: NCT04691947
Title: Phase 1 Study for the Determination of Safety and Immunogenicity of Two Different Strengths of the Inactivated COVID-19 Vaccine ERUCOV-VAC, Given Twice Intramuscularly to Healthy Volunteers, in a Placebo Controlled Study Design.
Brief Title: Safety and Immunogenicity of Two Different Strengths of the Inactivated COVID-19 Vaccine ERUCOV-VAC
Acronym: ERUCOV-VAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Health Institutes of Turkey (Other Government)
Collaborators: TC Erciyes University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IDEAL00420-EU01-PK537-1
Record Dates: First submitted 2020-11-14; First posted 2020-12-31 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: COVID-19 Vaccine
Keywords: COVID-19; Inactive Vaccine; Phase I
MeSH Terms: conditions — COVID-19 | interventions — TURKOVAC

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose vaccine (Experimental): Type: Biological/Vaccine Name: ERUCOV-VAC 3 µg/0.5 ml Vaccine Intervention Description:Two applications on Days 0 and 21
  Interventions: Biological: ERUCOV-VAC
- Medium dose vaccine (Experimental): Type: Biological/Vaccine Name: ERUCOV-VAC 6 µg/0.5 ml Vaccine Intervention Description: Two applications on Days 0 and 21
  Interventions: Biological: ERUCOV-VAC
- Placebo (Placebo Comparator): Placebo Vaccine, containing 0.9 % saline Intervention Description: Two applications on Days 0 and 21
  Interventions: Other: Placebo Vaccine

INTERVENTIONS:
Biological: ERUCOV-VAC — Vaccination on Day 0 and Day 21
  Arms: Low dose vaccine; Medium dose vaccine
Other: Placebo Vaccine — Placebo Vaccination on Day 0 and Day 21
  Arms: Placebo

SUMMARY:
The objective is to determine the safety and immunogenicity of two different strengths (3 µg and 6 µg) of an inactivated COVID 19 Vaccine compared to placebo so that to demonstrate the safety and efficacy in prophylaxis of COVID-19.

DETAILED DESCRIPTION:
This is a double-blind, double dose, parallel, randomized vaccination study. Each subject will receive in random order a double intramuscular dose of ERUCOV-VAC 3 µg/0.5 ml Vaccine, ERUCOV-VAC 6 µg/0.5 ml Vaccine or 0.5 ml of placebo Vaccine according to a sequence determined by randomization, on Day 0 (1st vaccination) and Day 21 (2nd vaccination).In total 34 healthy subjects of both genders will be monitored for one year in total, after Day 43 the study will be unblinded and the volunteers who took placebo vaccine will be released from the study. The most important evaluation will be performed on Day 43 after the first vaccine dose.

ELIGIBILITY:
Inclusion Criteria:

* healthy Caucasian origin
* age between 18 and 55 years
* accepting not to participate in another COVID-19 vaccine study until the end of the study
* volunteers who do not plan to get a child in the next one year; the volunteer and the partner should use a reliable form of contraception (abstinence, condom, birth control implant, birth control pills used or IUD used by the partner) during the study for at least 1 year
* participants must refrain from blood or plasma donation from the time of first vaccination until 3 months after last vaccination
* the outcome of the following examinations should be clinically insignificant: medical and surgical history (hypo-, hypertension, allergy, other diseases, major surgery, micturition, defecation, sleep, illness within the last 4 weeks prior to the start of the trial);
* life style and habits (consumption of alcohol, nicotine, coffee, tea, coke, special diet, drug abuse) should be normal/acceptable
* body temperature, pulse rate, blood pressure, respiratory rate and 12 lead ECG should be normal/acceptable.
* physical examination (general state and abnormal findings per system: endocrine/metabolic, allergies, drug sensitivities, head, neck, eyes, ears, nose, throat, cardiovascular, respiratory, gastrointestinal, hepatic/biliary, urogenital, musculoskeletal, lymph nodes, skin, and neurological/psychiatric) should be normal/acceptable
* laboratory examination (blood/serum examination: sodium, potassium, calcium, chloride, total protein, albumin, glucose, creatinine, BUN, uric acid, total bilirubin, direct and indirect bilirubin, lipid panel (total cholesterol, triglyceride, HDL, LDL), AST, ALT, GGT, ALP, haemoglobin, haematocrit, erythrocytes, leukocytes, platelet count, prothrombin time (PT) and activated partial thromboplastin time (aPTT); HBsAg, HIV-Ab, HCV-Ab; urine examination: urine color, appearance, specific gravity, pH, protein, glucose, ketones, blood, leukocytes, bilirubin, urobilinogen, nitrites and sediment if erythrocytes or leukocytes are out of the limits ) should be normal/acceptable.
* antiSARS CoV 2 total antibody (including COVID-19 IgG and/or IgM) negative in serum.
* drug screening negative (amphetamines, cannabinoids, benzodiazepines, cocaine, opioids, barbiturates)
* normal body weight in relation to height and age according to BMI (accepted range 18.5 and 30 kg/m2)

Exclusion Criteria:

* women with a positive blood (β-HCG) pregnancy test
* lactating women
* history of COVID-19 infection or showing COVID-19 infection symptoms
* having had contact to people with known COVID-19 infection in the last 14 days
* having fever (> 37.4oC in the last 24 hours), dry cough or feeling tired and having aches and pains, nasal congestion, runny nose, sore throat and diarrhea.
* positive real time RT-PCR COVID-19 test.
* persons with autoimmune diseases
* allergic diathesis or any clinically significant allergic disease (i.e. asthma)
* any condition that might impair the immune response
* recent or current immunosuppressive medication
* any other vaccine application 30 days before the first dose

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Non-pregnant women
Enrollment: 44 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of the COVID-19 vaccine | 43 days
  The number and proportion of subjects with adverse events observed until Day 43 post 1st vaccination are declared to be primary target variables.

SECONDARY OUTCOMES:
Serum IgG antibody Levels | 12 months
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s).
Neutralizing Antibodies Levels | 12 months
  Serum Neutralizing antibody levels.
TNF-alpha Levels | 12 months
  Serum TNF-alpha levels.
Interferon Levels | 12 months
  Serum IFN-γ levels.
Interleukine Levels | 12 months
  Serum IL-2, -4, -5, -6 levels.

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Sezer, Principal Investigator — Erciyes University Hakan Çetinsaya Iyi Klinik Uygulama ve Arastirma Merkezi, IKUM (Center for GCP)
Locations (1):
- Erciyes University Hakan Çetinsaya Iyi Klinik Uygulama ve Arastirma Merkezi, IKUM (Center for GCP), Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ozdarendeli A, Sezer Z, Pavel STI, Inal A, Yetiskin H, Kaplan B, Uygut MA, Bayram A, Mazicioglu M, Unuvar GK, Yuce ZT, Aydin G, Aslan AF, Kaya RK, Koc RC, Ates I, Kara A. Safety and immunogenicity of an inactivated whole virion SARS-CoV-2 vaccine, TURKOVAC, in healthy adults: Interim results from randomised, double-blind, placebo-controlled phase 1 and 2 trials. Vaccine. 2023 Jan 9;41(2):380-390. doi: 10.1016/j.vaccine.2022.10.093. Epub 2022 Nov 22. PMID 36460536